CLINICAL TRIAL: NCT07237763
Title: Comparison Between Topical Ketoconazole 2% Cream and Topical Adapalene 2% Cream in the Treatment of Mild Comedonal and Papulopustular Acne, a Randomized Controlled Trial
Brief Title: Assessment of the Efficacy of Topical Ketoconazole 2% Cream in Comparison With Topical Retinoids in the Treatment of Mild Comedonal and Papulopustular Acne
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mona Mostafa Korany Mahmoud, lecturer of dermatology, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dermatology 25
Record Dates: First submitted 2025-11-15; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Acne
Keywords: ketoconazole; adapalene
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mild acne patients who will apply topical ketoconazole 2% (Active Comparator): they will apply topical KTZ 2% cream twice daily on the whole face for 12 weeks
  Interventions: Drug: advised to apply topical ketoconazole 2% cream twice daily on the whole face.
- mild acne patients who will apply topical adapalene 2% (Active Comparator): they will apply topical retinoid cream once daily at night on the whole face except sensitive areas for a period of 12 weeks
  Interventions: Drug: topical adapalene to the face

INTERVENTIONS:
Drug: advised to apply topical ketoconazole 2% cream twice daily on the whole face. — ketoconazole will be applied twice per day on the face for 12 weeks
  Arms: mild acne patients who will apply topical ketoconazole 2%
Drug: topical adapalene to the face — will be advised to apply topical adapalene cream once daily at night on the whole face except sensitive areas for a period of 12 weeks
  Arms: mild acne patients who will apply topical adapalene 2%

SUMMARY:
objective: is to assess the efficacy of topical ketoconazole 2% cream in comparison with topical retinoid in the treatment of mild comedonal and papulopustular acne to determine if ketoconazole can be an alternative to topical retinoid with less side effects and more compliance.

Patients and methods: 52 patients with mild comedonal and papulopustular acne will be randomized into 2 groups and instructed to apply randomly either topical KTZ 2% cream or topical retinoid cream for a period of 12 weeks. Evaluation of response will be done by a blinded investigator

DETAILED DESCRIPTION:
Background: Acne vulgaris is a common chronic inflammatory skin disorder of pilosebaceous units that occurs predominantly in the skin of the face, upper chest and upper back. Acne is of multifactorial origin with four main pathophysiologic mechanisms: follicular hyperkeratinization with obstruction of pilosebaceous ducts, hormonal influences on sebum production, cutibacterium acnes (C. acnes) proliferation, immune host reaction and inflammation. Ketoconazole (KTZ) is an imidazolic anti-mycotic derivative that has been recently tried as a new line of treatment of mild acne. KTZ acts on microbial dysbiosis through the inhibitory effect on lipase activity of malassezia species and both antibiotic-susceptible and resistant C. acnes.

Objectives: our objective is to assess the efficacy of topical ketoconazole 2% cream in comparison with topical retinoid in the treatment of mild comedonal and papulopustular acne to determine if ketoconazole can be an alternative to topical retinoid with less side effects and more compliance.

Patients and methods: 52 patients with mild comedonal and papulopustular acne will be randomized into 2 groups. Group A will be advised to apply topical KTZ 2% cream twice daily on the whole face. Group B will be advised to apply topical retinoid cream once daily at night on the whole face except sensitive areas for a period of 12 weeks. Evaluation of response will be done by a blinded investigator 2 weeks after discontinuation of treatment using total lesion count, Global Evaluation of Acne (GEA) scores, Cardiff Acne Disability Index (CADI), and post-inflammatory hyperpigmentation (PIH) scores and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild comedonal or papulopustular acne with a GEA score from 1-2 on the face.
* Both sexes.
* Age: adolescents and adults.
* Skin type 3 and 4.

Exclusion Criteria:

* • Patients using, will use during the study, or discontinued less than 4 weeks before study baseline, prescribed or over-the counter topical therapies for the treatment of acne.

  * Patients using, will use during the study, or discontinued less than 4 weeks before study baseline, any facial procedures such as chemical peel, laser treatment or depilation in area of treatment application (except eyebrow shaping).
  * Patients with outdoor occupation, exposed to sun and heat.
  * Patients using, will use during study any cosmoceuticals.
  * Patients using, will use during the study, or discontinued less than 12 weeks before study baseline, systemic therapies for the treatment of acne or any other systemic treatments.
  * Patients with other special types of acne or conditions presenting with acne/acneiform eruption.
  * Irregular menstrual cycles or clinically suspected polycystic ovarian syndrome.
  * Patients with other facial rashes preventing the accurate assessment.
  * Known or suspected allergy to ingredients.
  * Pregnancy or lactation.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
To study the efficacy of topical ketoconazole 2% cream in treatment of mild to moderate acne | 3 months
  results will be assessed using total lesion count

SECONDARY OUTCOMES:
patient satisfaction | 3 months
  evaluation will be on a scale from 1-10
effect on post inflammatory hyperpigemntation | 3 month
  by a subjective score ranging from mild to severe

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes